CLINICAL TRIAL: NCT04364100
Title: Qualitative Study of the Experience of Hospital Students in the Odontology Department
Brief Title: Experience of Hospital Students in the Odontology Department
Acronym: EQUAVECU
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0255
Record Dates: First submitted 2020-03-09; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Occupational Stress
Keywords: Stress; well-being; anxiety; confidence; satisfaction
MeSH Terms: conditions — Occupational Stress; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During their studies, the dental students of Brest (France) learn their future profession by working in the Dental University Hospital, from the fourth academic year. This clinical activity is considered as both a source of satisfaction and stress by most of the students. The main objective of this study is to investigate the experience of Brest dental students through a qualitative methodology, with individual interviews, followed by an analysis by grounded theory (Paillé, 1994).

DETAILED DESCRIPTION:
During their studies, the dental students of Brest (France) learn their future profession by working in the Dental University Hospital, from the fourth academic year. This clinical activity is considered as a source of satisfaction by most of the students. They are also reassured because they know that they will easily find an employment at the end of their studies. However, the clinical activity can also create a stress among the students, which varies with their progress in their studies (Polychronopoulou et Divaris, 2009). Other sources of stress could also be identified. This multifactorial stress can influence their well-being, their practices and their relationships with patients. The stress and satisfactions of the dental students have mainly been studied by some questionnaires (Inquimbert et al., 2017). The main objective of this study is to investigate the experience of Brest dental students through a qualitative methodology, with individual interviews, followed by an analysis by grounded theory (Paillé, 1994). This type of research can enable us to keep a broad approach of students' experience and to stay faithful to it.

ELIGIBILITY:
Inclusion Criteria:

* volunteer students of Brest Dental University Hospital, having given his/her consent
* adult students of Brest Dental University Hospital, in fourth, fifth and sixth academic year

Exclusion Criteria:

* students in work-stoppage
* students in Erasmus program
* non-volunteer students or students refusing to give his/her consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer students of Brest Dental University Hospital in fourth, fifth and sixth academic year
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the hospital student (4th, 5th, 6th years) in odontology | 1 to 2 months
  Data collection until saturation: no new information after two consecutive interviews (theorizing)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Chevalier, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France